CLINICAL TRIAL: NCT03849872
Title: An Open-label, Single-dose Study to Evaluate the Excretion and Metabolism of Oral [14C]-ONO-5788 and Absolute Bioavailability of Oral ONO-5788 in Healthy Adult Male Subjects
Brief Title: Single-dose Study to Evaluate the Absolute Bioavailability and Mass Balance of ONO-5788
Acronym: ONO-5788-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-5788-02
Record Dates: First submitted 2019-02-14; First posted 2019-02-21 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Absolute Bioavailability (Experimental): Single oral dose of 10 mg ONO-5788 capsule followed by iv infusion 100 μg/ 41 kBq (1.1 μCi) [14C]-ONO-5788 in 6 healthy male subjects.
  Interventions: Drug: ONO-5788; Drug: [14C]-ONO-5788
- Part 2 Mass Balance (Experimental): Single oral dose of 10 mg [14C]-ONO-5788 capsule containing 4.1 MBq (111 μCi) [14C]-radioactivity in 6 healthy male subjects.
  Interventions: Drug: [14C]-ONO-5788

INTERVENTIONS:
Drug: ONO-5788 — Investigational Drug
  Arms: Part 1 Absolute Bioavailability
Drug: [14C]-ONO-5788 — Investigational Drug

SUMMARY:
A phase 1 healthy volunteer study to assess the excretion and metabolism as well as the absolute bioavailability of oral ONO-5788. The study will be conducted in two parts: Part 1 to assess the absolute bioavailability using ONO-5788 and radiolabelled ONO-5788 as intravenous and oral forms; part 2 will assess the mass balance of ONO-5788 using orally administered radiolabelled ONO-5788

ELIGIBILITY:
Inclusion Criteria:

1. The subject is willing and able to provide written informed consent.
2. Male subjects aged 21 to 65 inclusive at the time of signing the informed consent form.
3. The subject is able to communicate with the Investigator and the site staff.
4. A subject is eligible to participate if he is not trying to father a child, is willing to use one of the contraception methods listed in Section 5.3 and agrees not to donate sperm, from Day 1 of the study until 90 days after dosing.
5. The subject has a body mass index of 18.5 to 30.0 kg/m2, inclusive at screening.
6. The subject is healthy as determined by the Investigator (or medically qualified designee) based on the screening examinations including:

   * Medical history
   * Physical examination
   * Vital signs
   * 12-lead ECG
   * Clinical laboratory tests

   If any of the results of the above examinations are outside the locally-defined normal ranges, then the Investigator must consult with the Sponsor's Medical Officer prior to the subject being included in the study. Such subjects must only be included if the Investigator and Sponsor's Medical Officer believe the finding is unlikely to introduce additional risk for the subject if they enter the study.
7. The subject is a continuous non-smoker or has not used nicotine-containing products for at least 3 months prior to the first dose of study medication and will not use nicotine-containing products throughout the study, based on subject self-reporting.

Exclusion Criteria:

1. The Investigator deems the subject unsuitable for the study as a result of the screening examinations.
2. The subject is an employee of the Sponsor or contract research organization.
3. The subject has, or has a history of, any significant disease or disorder that would increase the risk for the subject if they were enrolled in the study or would affect study procedures or outcomes such as:

   1. Gallstones, cholangitis, and/or cholecystitis;
   2. Pancreatitis;
   3. Hypothyroidism;
   4. Known diabetes mellitus type 1 or type 2;
   5. Hypocalcaemia or hypokalaemia;
   6. Hypoglycaemia or hyperglycaemia or fasting blood glucose outside normal local range;
   7. Thrombocytopenia or other clinically significant haematologic abnormalities;
   8. Inflammatory bowel disease, irritable bowel syndrome, or abdominal surgery (with the exception of appendectomy);
4. The subject has a positive, pre-study, hepatitis B, hepatitis C or human immunodeficiency virus test.
5. The subject has clinically significant serum electrolyte (sodium, potassium, chloride, bicarbonate) abnormalities at screening or admission, in the estimation and clinical judgment of the Investigator or designee.
6. The subject has a history of regular alcohol use, within the previous 12 months, of >21 units/week. A unit is defined as a half-pint (240 mL) of beer, a small glass (125 mL) of wine or a single measure (25 mL) of spirits.
7. The subject has a supine blood pressure less than 90/40 millimeter of mercury (mmHg) or greater than 140/90 mmHg or a supine pulse rate lower than 50 beats per minute (bpm) or higher than 100 bpm at screening.
8. The subject has a history of regular use of drugs of abuse, including cannabinoids, cocaine, benzodiazepines, opioids, amphetamines, barbiturates, or methamphetamines within 1 year prior to first dose. Subjects who have been prescribed these drugs may be enrolled at the Investigator's discretion.
9. Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) at screening and (first) admission to the clinical research centre.
10. The subject has participated in a clinical trial within 3 months of dosing.
11. The subject has participated in more than 3 other drug studies in the 10 months prior to the first dose of study drug.
12. The subject has donated blood or had significant blood loss within 2 months prior to the first dose of study drug or has donated plasma within 7 days prior to the first dose of study drug.
13. The subject has used prescription medicine, non-prescription medicine, vitamins, herbal treatments or dietary supplements within 14 days of the first dose, unless in the opinion of the Investigator and Sponsor Medical Officer, the substance will not affect subject safety or interfere with the study procedures.
14. The subject has used any drugs known to be significant inducers or inhibitors of CYP enzymes and/or P-glycoprotein, including St. John's Wort, for 28 days prior to the first dose of study drug and throughout the study. Appropriate sources will be consulted by the Investigator or designee to confirm lack of interaction with study drugs.
15. The subject has a history of sensitivity to the study medication or the study medication class or any other drug.
16. The subject has an allergy that the Investigator or designee thinks may affect their safety during the study.
17. The subject is mentally or legally incapacitated.
18. The subject has been involved in a previous trial with ONO-5788.
19. The subject had a significant and/or acute illness within 5 days prior to dosing that, in the opinion of the Investigator, might impact safety assessments.
20. The subject has unsuitable veins for infusion or blood sampling.
21. The subject was exposed to radiation for diagnostic reasons (except dental xrays and plain xrays of thorax and bony skeleton [excluding spinal column]), during work, or during participation in a clinical study in the period of 1 year prior to screening.
22. The subject participated in another study with a radiation burden of >0.1 mSv and ≤1 mSv in the period of 1 year prior to screening; a radiation burden of >1.1 mSv and ≤2 mSv in the period of 2 years prior to screening; a radiation burden of >2.1 mSv and ≤3 mSv in the period of 3 years prior to screening, etc. (add 1 year per 1 mSv).
23. Part 2 only: The subject has an irregular defecation pattern (less than once per 2 days or clinically abnormal number of stools per day).

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male subjects only
Enrollment: 12 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability of ONO-5788 in plasma | 72 hours
  Absolute bioavailability is calculated from the AUCs of iv and oral administration
Mass balance of ONO-5788 | up to 42 days (until >90% of dose is recovered)
  Total recovery of radioactivity in urine and faeces following a single oral dose of [14C]-ONO-5788 (expressed as a percentage of the total radioactive dose administered)

SECONDARY OUTCOMES:
Pharmacokinetics (AUC) | Part 1: 24 hours through to 72 hours. Part 2: Day 1 to day 42 (depending on recovery of dose)
  Assessment of the plasma area under the curve of ONO-5788 and [14C]-ONO-5788
Pharmacokinetics (t1/2) | Part 1: 24 hours through to 72 hours. Part 2: Day 1 to day 42 (depending on recovery of dose)
  Assessment of the total elimination half life of ONO-5788 and [14C]-ONO-5788
Pharmacokinetics (CL) | 24 hours through to 72 hours.
  Assessment of the clearance of ONO-5788 (Part 1 only)
Pharmacokinetics (CL/F) | Part 1: 24 hours through to 72 hours. Part 2: Day 1 to day 42 (depending on recovery of dose)
  Assessment of Apparent oral clearance of ONO-5788
Pharmacokinetics (Vz) | 24 hours through to 72 hours.
  Assessment of Volume of distribution at terminal phase (Part 1 only)
Pharmacokinetics (Vz/F) | Part 1: 24 hours through to 72 hours. Part 2: Day 1 to day 42 (depending on recovery of dose)
  Assessment of Apparent volume of distribution at terminal phase
Pharmacokinetics (CLr) | Part 2: Day 1 to day 42 (depending on recovery of dose)
  Assessment of renal clearance (Part 2 only)
Treatment emergent adverse events | Part 1: 24 hours through to 72 hours. Part 2: Day 1 to day 42 (depending on recovery of dose)
  Number of participants with treatment emergent adverse events by severity
Clinical laboratory abnormalities | Part 1: 24 hours through to 72 hours. Part 2: Day 1 to day 42 (depending on recovery of dose)
  Number of participants with abnormalities in clinical laboratory results
Changes in vital signs | Part 1: 24 hours through to 72 hours. Part 2: Day 1 to day 42 (depending on recovery of dose)
  Number of participants with clinically significant changes in vital signs including pulse/heart rate, respiratory rate and blood pressure.
ECG abnormalities | Part 1: 24 hours through to 72 hours. Part 2: Day 1 to day 42 (depending on recovery of dose)
  Number of participants with ECG abnormalities
Physical examination assessment | Part 1: 24 hours through to 72 hours. Part 2: Day 1 to day 42 (depending on recovery of dose)
  A complete physical examination consisting of all body systems (except for genitalia and anus/rectal examinations, which will only be performed if medically indicated). Number of participants with clinically significant changes will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jaap van Lier, MD, Principal Investigator — PRA-EDS
Locations (1):
- PRA-EDS, Groningen, NZ, Netherlands